CLINICAL TRIAL: NCT00047554
Title: A Five-Year, Multicenter, Commercial Label Safety Study of TRAVATAN® 0.004% in Patients With TRAVATAN-Induced Iris Pigmentation Changes
Brief Title: Study of TRAVATAN in Subjects With Iris Pigmentation Changes
Status: Terminated | Type: Observational
Why Stopped: Study objectives met
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: C-01-79
Record Dates: First submitted 2002-10-08; First posted 2002-10-18 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension; primary open-angle glaucoma; iris; pigmentation
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — Travoprost; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- TRAVATAN: Travoprost, 0.004% ophthalmic solution, 1 drop to the study eye once daily in the evening for up to 5 years
  Interventions: Drug: Travoprost, 0.004% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost, 0.004% ophthalmic solution
  Other Names: TRAVATAN®

SUMMARY:
The purpose of this study was to monitor iris pigmentation changes over a 5-year period in patients with open-angle glaucoma or ocular hypertension. To be eligible for the study, these individuals must have experienced an iris pigmentation change while previously dosing with TRAVATAN.

ELIGIBILITY:
Inclusion:

* Diagnosis of open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component) or ocular hypertension;
* Has experienced an iris pigmentation change while dosing with TRAVATAN;
* Currently dosing with TRAVATAN;
* Other protocol-defined inclusion criteria may apply.

Exclusion:

* Any form of glaucoma other than open-angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component) or ocular hypertension;
* Not currently using TRAVATAN;
* Females of childbearing potential if pregnant, breast-feeding, or not using highly effective birth control measures;
* History of any severe ocular pathology (including severe dry eye);
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were identified and enrolled from 23 investigational centers in the US.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2003-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Iris Pigmentation from Baseline for Study Eye by Visit | Baseline, Up to Year 5
  As assessed by ocular photography

SECONDARY OUTCOMES:
Incidence of Change in Eyelash Characteristic from Baseline for Study Eye by Visit | Baseline, Up to Year 5
  As assessed by ocular photography

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, PhD, Study Director — Alcon Research